CLINICAL TRIAL: NCT00923598
Title: Optimizing Local Anesthetic Concentration for Continuous Femoral Nerve Blocks
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Brian M. Ilfeld, MD, MS, Associate Professor, In Residence, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Cleveland TKA Study
Record Dates: First submitted 2009-06-17; First posted 2009-06-18 (Estimated); Results first posted 2019-12-02 (Actual); Last update posted 2019-12-02 (Actual); Status verified 2019-11

CONDITIONS: Total Knee Arthroplasty; Knee Pain
Keywords: TKA; Bilateral; Cleveland Clinic; UCSD; Catheter; Nerve block; Postoperative pain; Femoral Catheter; Bilateral Total Knee Arthroplasty; Bilateral Femoral Catheter
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1) 0.1% Ropivicaine on Right Leg (Active Comparator): Patients will be randomized ot 0.1% Ropivicaine infusion on the right leg and therefore 0.4% Ropivicain in fusion for the left leg for pain due to bilateral TKA. The outcome measures will be measured on both legs, starting with the right leg each time. The infusion will last for the two days following surgery, that the patient is staying in the hospital.
  Interventions: Drug: 0.1% and 0.4% perineural ropivicaine
- 2) 0.4% Ropivicaine on Right Leg (Active Comparator): Patients will be randomized ot 0.4% Ropivicaine infusion on the right leg and therefore 0.1% Ropivicain in fusion for the left leg for pain due to bilateral TKA. The outcome measures will be measured on both legs, starting with the right leg each time. The infusion will last for the two days following surgery, that the patient is staying in the hospital.
  Interventions: Drug: 0.1% and 0.4% perineural ropivicaine

INTERVENTIONS:
Drug: 0.1% and 0.4% perineural ropivicaine — Patients will be randomized to one of two groups: Ropivicaine 0.1% infusion on the right leg and Ropivicaine 0.4% infusion on the left leg, or Ropivicaine 0.4% infusion on the right leg and Ropiviciane 0.1% infusion on the left leg for treatment of postoperative pain following bilateral TKA. Both groups will receive the same total dose of medication and will have the infusion for the two days following surgery.

SUMMARY:
This is a randomized, observer-masked, controlled study. Subjects will be patients undergoing bilateral total knee arthroplasty (TKA). One side (left or right) will be randomized to one of two treatment groups: a postoperative ropivacaine concentration of 0.1% or 0.4%. The contralateral side will receive the other possible ropivacaine concentration of 0.1% or 0.4%. The basal rate and patient-controlled bolus volume will depend upon the treatment group, but the total dose of local anesthetic is the same for each. For the duration of the study, all patients will receive the current usual and customary analgesics for bilateral TKA patients. All patients will receive a ropivacaine perineural infusions initiated in the operating room and continued until at least the afternoon of postoperative day (POD) 2, as well as oral acetaminophen, a sustained-release oral opioid; and celecoxib. Rescue opioid and route of administration will be determined by pain severity using a Numeric Rating Scale of 0-10, with 0 equal to no pain and 10 being the worst imaginable pain.

DETAILED DESCRIPTION:
The investigators propose to test the null hypothesis that differing concentrations of ropivacaine (0.1% vs. 0.4%) at an equal total dose has no impact on quadriceps muscle strength during a continuous femoral nerve block following total knee arthroplasty (TKA). These results will help define the optimal concentration of local anesthetic used for continuous peripheral nerve blocks.

ELIGIBILITY:
Inclusion Criteria:

* Primary, bilateral TKA
* Age 18 years or older
* Postoperative analgesic pain includes bilateral continuous femoral nerve blocks

Exclusion Criteria:

* Chronic, high-dose opioid use
* History of opioid abuse
* Any neuro-muscular deficit of either femoral nerves and/or quadriceps muscles
* Pregnancy
* Incarceration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2009-06; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel I Sessler, M.D., Principal Investigator — The Cleveland Clinic, Chair, Department of Outcomes Research
Locations (1):
- The Cleveland Clinic, Main Campus, Cleveland, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 1) 0.1% Ropivicaine on Right Leg | 2) 0.4% Ropivicaine on Right Leg
Started | 23 | 22
Completed | 19 | 17
Not Completed | 4 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 1) 0.1% Ropivicaine on Right Leg | 2) 0.4% Ropivicaine on Right Leg | Total
Number analyzed (Participants) | 23 | 22 | 45
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 18 | 11 | 29
  >=65 years | 5 | 11 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 60 (9) | 60 (9) | 60 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 11 | 21
  Male | 13 | 11 | 24
Region of Enrollment [Number; unit: participants]
  United States | 23 | 22 | 45

OUTCOME MEASURES:

1. Primary Outcome: Quadriceps Femoris Muscle Strength Maximum Voluntary Isometric Contraction (MVIC)
Description: A device was used called a dynamometer to measure the force during maximum voluntary isometric contraction. The dynamometer was placed on ipsilateral anterior tibia perpendicular to the tibial crest, just proximal to the medial malleolus. Subjects were asked to take 2 seconds to come to maximum effort contracting the quadriceps, maintain this effort for 5 seconds, and then relax.
Time Frame: morning of postoperative day 2
Population: Patients undergoing bilateral knee replacements
Measure: Mean (Standard Deviation); unit: newtons
Arm/Group | 1) 0.1% Ropivicaine on Right Leg | 2) 0.4% Ropivicaine on Right Leg
Number analyzed (Participants) | 23 | 22
newtons | 13 (8) | 12 (8)
Statistical Analysis 1: Comparison: 1) 0.1% Ropivicaine on Right Leg vs 2) 0.4% Ropivicaine on Right Leg; Test type: Equivalence — A method by Armitage et al was used, where by equivalence of treatments would be concluded if the 95% CI for the difference fell within the prespecified tolerated interval. Under these assumptions, a trial with 36 subjects (72 limbs) would correctly conclude there is no treatment difference with probability 80%, and incorrectly conclude equivalence when there is a difference of 20% with probability 5%; p = 0.05, Fisher Exact; Mean Difference (Final Values) = 3, 95% CI 2-sided [-10 to 17]

ADVERSE EVENTS:
Arm/Group | 1) 0.1% Ropivicaine on Right Leg | 2) 0.4% Ropivicaine on Right Leg
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/22
Other Adverse Events (participants affected / at risk) | 0/23 | 0/22

LIMITATIONS AND CAVEATS:
Study may not be applicable to other catheter designs or insertion techniques; local anesthetic types, concentrations, or doses; infusion delivery methods or durations; and certainly anatomic catheter locations.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes